CLINICAL TRIAL: NCT06531460
Title: Effect of Perioperative Nutrition Enriched With Omega-3 on the Incidence of Infections in Oncologic Patients Following Lung Resection
Brief Title: Nutritional Therapy Enriched With Omega-3 in Patients With Lung Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Ivan Armando Osuna Padilla, Clinical Nutrition Manager, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C34-24
Record Dates: First submitted 2024-07-26; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Surgery
Keywords: lung cancer; omega-3; prehabilitation nutrition; perioperative nutrition; infections; inflammation response
MeSH Terms: conditions — Lung Neoplasms; Infections | interventions — Enteral Nutrition; Fish Oils; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Use of enteral formula enriched with omega-3 or standard not revealed for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental enteral nutrition (Experimental): Patients admitted to the hospital at least three days before surgery Use of an enteral feeding tube to administer enriched enteral formula
  Interventions: Dietary Supplement: Fish oil enteral supplementation
- Experimental oral nutrition (Experimental): Patients admitted one day before surgery. Home-self administration of enriched enteral formula three days before surgery
  Interventions: Dietary Supplement: Fish oil oral supplementation
- Standard enteral nutrition (Other): Patients admitted to the hospital at least three days before surgery Use of an enteral feeding tube to administer standard enteral formula
  Interventions: Dietary Supplement: Enteral nutrition without fish oil
- Standard oral nutrition (Other): Patients admitted one day before surgery. Home-self administration of standard enteral formula three days before surgery
  Interventions: Dietary Supplement: Oral nutritional supplement without fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil enteral supplementation — Omega-3 (4.2 g), administered through an enteral feeding tube, three days before surgery
  Arms: Experimental enteral nutrition
Dietary Supplement: Fish oil oral supplementation — Omega-3 (4.2 g), orally administered enriched nutritional formula, drinking at home three days before surgery
  Arms: Experimental oral nutrition
Dietary Supplement: Enteral nutrition without fish oil — Enteral formula without omega-3 administered through an enteral feeding tube, three days before surgery
  Arms: Standard enteral nutrition
Dietary Supplement: Oral nutritional supplement without fish oil — Oral nutritional supplement without omega-3 orally administered, drinking at home three days before surgery
  Arms: Standard oral nutrition

SUMMARY:
The aim of this study is to analyze the effect of enriched formula with omega-3 in the 30-day incidence infection and inflammatory response following lung resection surgery in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer diagnosis
* Elective surgery for lung resection schedule at least four days before surgery
* Signed informed consent.

Exclusion Criteria:

* Acute or chronic organ failure as hepatic or renal insufficiency
* Patients with fish-allergy
* History of any surgery within 3 months
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
30-day incidence infection | 30-day incidence infection following lung resection in lung cancer patients.
  Incidence of infectious complications after surgery diagnosed using any of these criteria:
  Infection of surgery wound confirmed by culture Infection confirmed by blood culture Pneumonia developed after surgery confirmed by chest x Ray.

SECONDARY OUTCOMES:
Changes in prostaglandin E2 | At the beginning of nutritional therapy and at day-4 following surgery
  Measured in serum sample made by Enzyme-linked immunosorbent assay (ELISA).
Changes in Interleukin-6 | At the beginning of nutritional therapy and at day-4 following surgery
  Measured in serum sample made by Enzyme-linked immunosorbent assay (ELISA).
Changes in Tumor Necrosis Factor Alpha (TNF-α) | At the beginning of nutritional therapy and at day-4 following surgery
  Measured in serum sample made by Enzyme-linked immunosorbent assay (ELISA).
Number of participants with therapeutic antibiotics prescription | During the hospital stay until 30-day
  Frequency of therapeutic antibiotics prescription will be collected from medical records and medication administration registers.
Hospital lenght of stay | During the hospital stay until 90-day
  Number of calendar days that elapsed since hospital admission to the day of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ivan A Osuna-Padilla, PhD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No